CLINICAL TRIAL: NCT01043718
Title: Delivering an Evidence-Based Lifestyle Intervention Via the Internet: A Randomized Controlled Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Milton S. Hershey Medical Center (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen McTigue, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMC32877
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Obesity; Internet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- More-Intensive (Experimental)
  Interventions: Behavioral: More-Intensive
- Less-Intensive (Active Comparator)
  Interventions: Behavioral: Less-Intensive

INTERVENTIONS:
Behavioral: More-Intensive — The online lifestyle intervention will include elements of a behavioral lifestyle program developed by the Diabetes Prevention Program. The program will assist individual participants with establishing appropriate weight loss goals, implementing dietary recommendations (including analysis of current diet), and defining exercise programs. The program curriculum provides standard information about healthy lifestyle, and behavioral techniques for integrating them into daily living. In each lesson, patients provide feedback about how they interpret the information, and ideas for integrating it into their lives.
  Arms: More-Intensive
Behavioral: Less-Intensive — The participants will be provided with the information to access the online Diabetes Prevention Program (DPP) intervention materials. Following the original DPP trial, all DPP materials were placed online for the public to access. This group will receive a lifestyle counseling session and tools to facilitate their intervention.
  Arms: Less-Intensive

SUMMARY:
Hershey Medical Center and the University of Pittsburgh are doing a research study to help meet the needs of the adult population at risk for diabetes and heart disease. This study will provide a web-based program that aims to help participants to develop healthier eating habits, lose weight and become more physically active. The Internet-based materials will teach participants about healthy eating and physical activity and will ask them to incorporate the information they learn into their daily lives.

The purpose of this study is to evaluate the effectiveness of online lifestyle change programs to promote weight loss, healthy eating and physical activity patterns, in the interest of reducing risk for and adverse outcomes of type 2 diabetes (T2D) and cardiovascular disease (CVD).

ELIGIBILITY:
Please note: Only individuals who receive primary care at one of the Internal Medicine clinics at Milton S. Hershey Medical Center in Hershey, PA, are eligible for this study.

Inclusion Criteria:

* Age between 18 and 80 years old
* Obese based on World Health Organization criteria (BMI>30kg/m2)
* Receiving primary care from and referred by a provider at one of the Internal Medicine clinics at Milton S. Hershey Medical Center in Hershey, PA
* Able to understand and sign an informed consent document
* Able to communicate with the investigator and understand the requirements of this study

Exclusion Criteria

* Primary care provider determines that the individual is unable to safely undertake moderately intense unsupervised physical activity (the equivalent of 30 minutes of brisk walking)
* Primary care provider determines that the individual has inadequate cognitive function to participate in either active intervention curricula
* Women who are pregnant, who are planning to become pregnant in the next two years, or who become pregnant during the study
* Women who are breastfeeding
* Prisoners
* Children
* Individuals who are planning to have bariatric surgery or who have had bariatric surgery in the past two years
* Individuals with uncontrolled hypertension (systolic blood pressure (SBP) >165, diastolic blood pressure (DBP) >100)
* Individuals with an edematous state that interferes with body weight assessment (e.g., severe congestive heart failure, end- stage renal disease, or ascites),
* Individuals already using weight loss therapy
* Individuals with an inability to learn adequately from English language audio-taped materials
* Individuals with a lack of high-speed Internet access (Internet access will be based on participant perception; for example, participants could use computers belonging to friends, relatives, or libraries if they feel that they can access them regularly)
* Individuals without access to a scale
* Individuals unable to attend an Orientation session at Hershey Medical Center in Hershey, PA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | 6 months, 12 months, 18 months

SECONDARY OUTCOMES:
Percentage of body weight lost | 6 months, 12 months, 18 months
Change in blood pressure (mm Hg) | 6 months, 12 months, 18 months
Change in health-related quality of life as determined by the RAND-36 PCS or MCS | 6 months, 12 months, 18 months
Change in physical activity (steps per day) | 6 months, 12 months, 18 months
Change in dietary pattern | 6 months, 12 months, 18 months
Satisfaction with program | 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen McTigue, MD MS MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955